CLINICAL TRIAL: NCT00543985
Title: Exercise in Patients With Metabolic Syndrome and Weight Regain - Echocardiography Substudy
Brief Title: Exercise,Metabolic Syndrome and Weight Regain (Echocardiography Substudy)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R01DK067036 (Echo substudy); R01DK067036 (NIH)
Record Dates: First submitted 2007-10-11; First posted 2007-10-15 (Estimated); Results first posted 2016-11-22 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2016-11

CONDITIONS: Metabolic Syndrome; Obesity
Keywords: metabolic syndrome; obesity; exercise
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stress Echocardiography (Experimental): Echocardiography was performed prior to and within 60 seconds of completing the standard Bruce treadmill protocol.
  Interventions: Procedure: Stress Echocardiography

INTERVENTIONS:
Procedure: Stress Echocardiography — Echocardiography was performs prior to and within 60 seconds of completing the standard Bruce treadmill protocol.

SUMMARY:
We plan to test the hypothesis that patients with metabolic syndrome will have impaired left ventricular diastolic parameters. These parameters will be measured before and after a stress test at the end of a 3 month period of exercise training and a 10% weight loss.

DETAILED DESCRIPTION:
Patients must have 2 of the 5 criteria for metabolic syndrome and be able to exercise in a monitored setting for 45 min 5 times a week.

ELIGIBILITY:
Inclusion Criteria:

* 2 of 5 criteria for metabolic syndrome
* Ability to exercise for 45 min 5 days a week

Exclusion Criteria:

* No diabetes
* Established coronary disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom R Thomas, PhD, Principal Investigator — University of Missouri-Columbia; Kevin C Dellsperger, MD, PhD, Study Director — University of Missouri-Columbia; Anand Chockalingam, MD, Study Director — University of Missouri-Columbia

REFERENCES:
- [Result] Chockalingam A, Linden MA, Dellsperger KC, Thomas TR. Correlation of Normal Diastolic Cardiac Function With VO in the Metabolic Syndrome. Prev Cardiol. 2009 Summer;12(3):163-8. doi: 10.1111/j.1751-7141.2009.00027.x. PMID 19523060

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited as part of the parent study on Weight Regain (PI Tom Thomas) funded by NIH. These patients were recruited from clinics, volunteers from advertisements. Patients needed to have 2 of 5 criteria for the Metabolic Syndrome (MetS) plus have obesity.
Pre-assignment Details: All patients in this study had successfully been screened as part of the parent study. All patients were to exercise (aerobic) and have a 10% weight loss. Echocardiography was performed prior to and immediately following a maximal stress test at the end of 12 weeks of exercise.
Period: Overall Study
Arm/Group | Stress Echocardiography
Started | 36
Completed | 32
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Groups:
- Stress Echocardiography: Patients completed 3 months of training with 10% weight loss. At the end of that study, they were subjected to pre- and post-stress echocardiography to evaluate E/E' and VO2 max.
Arm/Group | Stress Echocardiography
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (2)
Gender [Count of Participants; unit: Participants]
  Female | 15
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Mean Resting E/E'
Description: E/E' is an echocardiographic parameter where E = early mitral inflow velocity and E' = early diastolic mitral annular motion. Measured in all participants prior to treadmill stress test.
Time Frame: 12 weeks
Population: The echo results from all subjects were analyzed at rest and following maximal exercise testing.
Measure: Mean (Standard Error); unit: ml/min/kg
Groups:
- Stress Echocardiography: Echocardiogram E/E' measured before and after exercise
Arm/Group | Stress Echocardiography
Number analyzed (Participants) | 32
ml/min/kg | 7.01 (0.37)
Statistical Analysis 1: Comparison: Stress Echocardiography; Pearson Product correlation was used to determine relationships between resting E/E' and Exercise VO2 max and Stress E/E' and Exercise VO2max; Test type: Superiority or Other; p = 0.14, Regression, Linear; Pearson correlation coefficient = -0.266

2. Primary Outcome: Post-exercise E/E'
Description: E/E' is an echocardiographic parameter where E = early mitral inflow velocity and E' = early diastolic mitral annular motion. Measured in all participants immediately following treadmill stress test.
Time Frame: 12 weeks
Population: The echo results from all subjects were analyzed at rest and following maximal exercise testing.
Measure: Mean (Standard Error); unit: ml/min/kg
Groups:
- Stress Echocardiography: Echocardiogram E/E' measured after exercise
Arm/Group | Stress Echocardiography
Number analyzed (Participants) | 32
ml/min/kg | 7.41 (0.41)

3. Secondary Outcome: Mean Resting Maximal Oxygen Uptake (VO2 Max)
Description: Measure of the maximum volume of oxygen that a body is capable of utilizing in one minute, measured in milliliters per kilogram of body weight per minute (ml/kg/min). Measured in all participants prior to treadmill stress test.
Time Frame: 12 weeks
Population: This data, if analyzed, is unavailable as the PI/study staff left the institution before completing the analysis and without making results available.
Arm/Group | Stress Echocardiography
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Maximal Oxygen Uptake (VO2 Max)
Description: Measure of the maximum volume of oxygen that a body is capable of utilizing in one minute, measured in milliliters per kilogram of body weight per minute (ml/kg/min) Measured in all participants immediately following treadmill stress test.
Time Frame: 12 weeks
Population: as for outcome 3
Arm/Group | Stress Echocardiography
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Stress Echocardiography: Patients completed 3 months of training with 10% weight loss. At the end of that study, they were subjected to pre- and post-stress echocardiography to evaluate E/E' .
Arm/Group | Stress Echocardiography
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No